CLINICAL TRIAL: NCT03907865
Title: Clinical Efficacy of Topical Hydrocortisone 0.335% (Softacort®) in Patients With Chronic Dry Eye Disease and Associated Ocular Surface Inflammation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: T1565-PIV-0117
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intense (Experimental): Patients have been randomized to receive Softacort eye drops for 12 days 4 times daily followed by 2 days twice daily treatment resulting in a total time of 14 days
  Interventions: Drug: Softacort
- standard (Experimental): Patients have been randomized to receive Softacort eye drops for 8 days 3 times daily followed by 3 days twice daily treatment resulting in a treatment time of 11 days total
  Interventions: Drug: Softacort

INTERVENTIONS:
Drug: Softacort — Group 1: 4 times daily for the first 12 days of the treatment period and then 2 times daily for 2 additional days Group 2: 3 times daily for the first 8 days of the treatment period and then 2 times daily for 3 additional days

SUMMARY:
Dry eye disease (DED) is a highly prevalent ocular condition and induces a significant burden to the affected patients. Regardless of the underlying etiology, DED is associated with increased inflammation of the entire ocular surface including the adnexa, conjunctiva and cornea. As such, there is evidence from in vitro, animal and clinical studies that this inflammatory response of the ocular surface plays a pathophysiological key role in the development of DED. The Dry Eye Workshop 2007 (DEWS) therefore suggests the use of anti-inflammatory drugs such as corticosteroids, cyclosporine or others when topical lubricants alone are not sufficient. Recently, Softacort® eye drops containing 0.335% hydrocortisone have gained marketing authorization for the treatment of ocular surface inflammation. This formulation offers several advantages that make them potentially interesting for the treatment of DED. First, the formulation is preservative-free, which is of special importance in patients with DED, since it has been shown that preservatives are detrimental for the ocular surface. Further, hydrocortisone has the advantage that in comparison to other glucocorticoid derivatives, it features poor solubility. This means that corneal penetration is low, which is a desired effect in the treatment of ocular surface inflammation. Because of the poor penetration through thecornea, elevation of intraocular pressure and cataract formation, which are common side effect of corticosteroid treatment, have not been observed with Softacort® to date, also favoring the use of this agent in DED. The aim of the present study is to investigate whether treatment with Softacort® improves ocular surface inflammation as well as clinical signs and symptoms associated with DED in patients who are already taking topical lubricants for at least three months.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years
* Normal ophthalmic findings except dry eye disease
* Ametropy ≤ 6 diopters
* Chronic dry eye defined as longer than six months since diagnosis
* OSDI ≥ 22
* Conjunctival Hyperemia ≥ Grade 3 (Efron Scale)
* Current use of topical lubricants since at least 3 months

Exclusion criteria:

* Best far corrected visual acuity < 1/10
* Severe Dry Eye associated with:
* Eyelid malposition
* Sjogren Syndrome
* Steven Johnson Syndrome
* Corneal dystrophy
* Ocular neoplasia
* Filamentous keratitis
* Corneal neovascularisation
* Orbital radiotherapy
* History of any of the following within last 3 months:
* Systemic treatment of dry eye
* Systemic treatment of MGD
* Isotretinoide,
* Cyclosporine,
* Tacrolimus, Siromilus, Pimecrolimus
* Punctual plugs
* Anti-glaucoma treatment
* History of any of the following within previous six months:
* ocular trauma
* ocular infection, ocular allergy
* History of any of the following within last 12 months:
* inflammatory corneal ulcer
* Herpetic eye infection or uveitis
* Ocular surgery
* History of IOP increase caused by systemic or topical treatment with corticosteroids
* IOP > 22mmHg
* Glaucoma in the medical history
* Known hypersensitivity to any of the components of the IMP under investigation or other study medication
* Allergic rhinitis; active or susceptible to reactivation during the study
* Pregnant or breast-feeding woman.
* Woman of childbearing potential (neither menopausal, nor hysterectomized, nor sterilized) not using effective contraception (oral contraceptives, intrauterine device, contraceptive implant or condoms)
* Inability of patient to understand the investigation procedures and thus inability to give valid, informed consent.
* Non-compliant patient (e.g. not willing to attend the follow-up visits, way of life interfering with compliance)
* Participation in another clinical study or clinical investigation at the same time as the present investigation
* Participation to the present clinical investigation during the exclusion period of another clinical study
* Patient already included once in this clinical investigation
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2019-01-02 (Actual)

PRIMARY OUTCOMES:
Conjunctival hyperemia | 5 minutes
  Conjunctival hyperemia will be graded according to the Efron Scale: 0=none, 1=trace, 2 = mild, 3 = moderate, 4 = severe

OTHER OUTCOMES:
Corneal fluorescein staining according to the Oxford Scale | 5 minutes
  Minims-Fluorescein Sodium 2.0% eye drops will be used to detect corneal epithelial defects. As grading scale for corneal damage, the NEI/Industry Workshop guidelines will be used 1. The cornea will be divided into five sectors (central, superior, inferior, nasal and temporal), each of which is scored on a scale of 0-3, whereas 0 means no staining and 3 means maximum staining, with a maximal score of 15.
  Corneal staining will also be graded according to the Oxford Scale (Annex II).
Tear film thickness | 30 minutes
  Tear film thickness as measured with ultra-high resolution optical coherence tomography (OCT)
Tear osmolarity | 5 minutes
  Tear film osmolarity will be measured non-invasive with a commercially available instrument (TearLab®, OcuSens Inc, San Diego, USA). The TearLab® technology uses an approach that concentrates laboratory functions on a single chip that requires less than 50 nL of tear fluid in order to measure tear osmolarity.
  The system uses a handheld pen on which the ophthalmologist places the noninvasive laboratory chip test card. Then the tear sample is collected by pressing the tip of the pen towards the conjunctiva adjacent to the lower lid margin. The collection of the tear sample takes usually less than 30 seconds and is painless for the subject.
HLA-DR expression | 20 minutes
  2 samples will be taken from the upper conjunctiva of the study eye using EYEPRIM™ (Opia Technologies S.A.S., Paris, France). The subject will be instructed to look down. The device will be positioned upon the conjunctiva. Then, the push-button will be pressed until the stop position is reached and then be held in this position for 2-3 seconds. Afterwards, the pressure will be released and the device will be removed from the eye. The sampling membrane will be ejected in a storage container by pressing the push-button once again. The samples will be stored according to the manufacturer's instructions and will be sent under observer blinded conditions to an independent laboratory (Iris Pharma, La Gaude, France) for analysis and assessment of HLA-DR levels.
Ocular surface disease index (OSDI©) | 5 minutes
  Symptoms of dry eye will be assessed using the Ocular Surface Disease Index© (OSDI©) which was developed by the Outcomes Research Group at Allergan Inc (Irvine, Calif)27. The questionnaire that underlies the OSDI© is specifically designed for patients with dry eye syndrome and asks patients about the frequency of specific symptoms and their impact on vision-related functioning. A sample of the OSDI© in German is given in Annex III.
Intraocular pressure | 5 minutes
  Intraocular pressure will be measured with a slit-lamp mounted Goldmann Applanation Tonometer.
  Before each measurement one drop of oxybuprocainhydrochloride combined with sodium fluorescein will be used for local anesthesia of the cornea.
Visual acuity | 5 minutes
  Best-corrected visual acuity will be measured using the standard ETDRS acuity charts.
Visual analogue scale (VAS) for patient satisfaction | 5 minutes
  Patient satisfaction assessed by a VAS will be determined using a 100 mm VAS on which 0 means "I do not agree" and 100 means "I totally agree". The following questions will be assessed using VAS: "I feel satisfied using this treatment" "With these eye drops, I have a feeling of freshness" "With these eye drops, I have a feeling of relief" "This product contributed to reduce my pain due to eye dryness" "This product is comfortable"

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University Vienna, Vienna, Austria

REFERENCES:
- [Derived] Kallab M, Szegedi S, Hommer N, Stegmann H, Kaya S, Werkmeister RM, Schmidl D, Schmetterer L, Garhofer G. Topical Low Dose Preservative-Free Hydrocortisone Reduces Signs and Symptoms in Patients with Chronic Dry Eye: A Randomized Clinical Trial. Adv Ther. 2020 Jan;37(1):329-341. doi: 10.1007/s12325-019-01137-8. Epub 2019 Nov 18. PMID 31741283